CLINICAL TRIAL: NCT07321392
Title: PSYCHOMETRIC VALIDATION OF THE PSYCHOSOCIAL ASSESSMENT TOOL IN CAREGIVERS OF PEDIATRIC CANCER PATIENTS.
Status: Active, not recruiting | Type: Observational
Sponsor: Aquí Nadie Se Rinde I.A.P. (Other)
Responsible Party: Principal Investigator, Alejandro Hernández Posadas, External researcher., Aquí Nadie Se Rinde I.A.P.
Other Study IDs: HIM-2023-049
Record Dates: First submitted 2025-12-09; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Patients With Cancer; Informal Primary Caregivers
Keywords: Neoplasms; Child; Caregivers; Psychometrics; Psychological Tests
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Psychosocial Assessment Tool (PAT) — The PAT is a brief report for informal primary caregivers that assesses family psychosocial risk based on a families' ecological social model. This model assesses psychosocial risks throughout the child's social environment and generates seven subscale scores, such as Family Structure/Resources, Social Support, Children's Problems, Sibling Problems, Family Problems, Stress Reactions, and Family Beliefs. The total score, which ranges from 0 to 7, is assigned to the PPPHM with three risk levels: universal (<1.00), specific (1.00 and 2.00) and clinical (>2.00). To translate the PAT into Spanish, methods that met or exceeded the guidelines of Holmbeck and Devine were used. First, the PAT was independently translated and back-translated by two native Spanish-speaking psychologists [62]. Then, an independent native Spanish speaker reviewed it and consulted with a certified translator.

SUMMARY:
The reported mental health, economic and structural problems of pediatric cancer patients end up negatively affecting family functioning and the course of the disease; therefore, in the Mexican context it is necessary to have a valid, reliable and culturally relevant tool to identify psychosocial risks in children and adolescents with cancer. in order to develop strategies to address psychosocial needs. Objective: To determine the psychometric validation of the Mexican version of the Psychosocial Assessment Tool (PAT) for informal primary caregivers of pediatric cancer patients. Method: A study will be carried out with a prospective multicenter instrumental design of correlational scope and a non-probabilistic sampling will be used at the convenience of informal primary caregivers of pediatric cancer patients. The indices of relevance, writing and adequate language will be evaluated, in order to obtain content validity of each of the 68 items, using the Aiken V, reliability will be evaluated by calculating the Kuder-Richardson 20 coefficient to determine internal consistency and structural or construct validity will be evaluated by means of an exploratory factor analysis. Results: According to the guidelines for adaptation and validation of psychological instruments, the inventory will be translated into the original language (English - Spanish), the inventory will be backtranslated into the original language (Spanish - English), the evidence of content validity will be obtained by expert judges, and the evidence of construct validity and reliability indices of the inventory will be piloted and obtained with the white sample.

Keywords: Pediatric patients, cancer, psychosocial risk, informal primary caregivers, pediatric oncology.

DETAILED DESCRIPTION:
In the Mexican context, it is necessary to have a valid, reliable and culturally relevant tool to identify psychosocial risks in children and adolescents with cancer, because, due to social, economic, cultural and psychological factors, these patients and their families are at risk, therefore, the validation of the psychosocial risk is not the same as theThe psychometric analysis of the Psychosocial Assessment Tool would allow an adequate diagnosis so that the multidisciplinary team can use interventions aimed at the specific needs of the patient and their relatives in multiple contexts where they work, regardless of the type of neoplasm or the phase of treatment in which they are.

Hypothesis

Statistical hypothesis:

Validation based on internal structure H1: r ≥ 0.7 H0: r < 0.7 Validation content-based H1: V ≥ 0.8 H0: V < 0.8

Methodological hypotheses:

Validation based on internal structure H1: There will be validation evidence based on the internal structure of the Psychosocial Assessment Tool (PAT) in its Mexican version for informal primary caregivers of pediatric cancer patients.

H0: There will be validation evidence based on the internal structure of the Psychosocial Assessment Tool (PAT) in its Mexican version for informal primary caregivers of pediatric cancer patients.

Content-based validation H1: There will be validation evidence based on the content of the Psychosocial Assessment Tool (PAT) in its Mexican version for informal primary caregivers of pediatric cancer patients.

H0: There will be validation evidence based on the content of the Psychosocial Assessment Tool (PAT) in its Mexican version for informal primary caregivers of pediatric cancer patients.

Research Question What will be the psychometric properties of the Psychosocial Assessment Tool (PAT) in its Mexican version for informal primary caregivers of pediatric cancer patients? General objective To determine the psychometric validation of the Mexican version of the Psychosocial Assessment Tool (PAT) for informal primary caregivers of pediatric cancer patients.

Specific objectives

* To translate the Psychosocial Assessment Tool (PAT) in its Spanish version for informal primary caregivers of Mexican pediatric cancer patients.
* To determine the content validity of the Spanish version of the Psychosocial Assessment Tool (PAT) for informal primary caregivers of Mexican pediatric cancer patients.
* To obtain the confirmatory factor structure of the Mexican version of the Psychosocial Assessment Tool (PAT) for informal primary caregivers of pediatric cancer patients.
* To estimate the internal consistency index of the Mexican version of the Psychosocial Assessment Tool (PAT) for informal primary caregivers of pediatric cancer patients.
* To obtain the exploratory factor structure of the Mexican version of the Psychosocial Assessment Tool (PAT) for informal primary caregivers of pediatric cancer patients.

Type of study It is a non-experimental , observational analytical, prospective, and multicenter analytical research design, since it is analytical because it quantifies the relationship between two factors, which are the effect of an intervention or an exposure, and observational because it is passive and does not modify the independent variables. It is transversal, since it examines the occurrence of a variable in a defined population at a particular time and prospective, since they begin with the observation of certain presumed causes and advance longitudinally in time in order to observe their consequences. Finally, it is multicenter because it will be conducted at more than one medical institution; for example, the present study will be conducted at the National Institute of Pediatrics and the Federico Gómez Children's Hospital of Mexico.

Design According to the characteristics of this study and the classification of research in clinical and health psychology [65], it is an instrumental design, because it is aimed at obtaining the psychometric properties of an inventory.

Identification and definition of variables In accordance with the main objective of the study, to validate the Psychosocial Assessment Tool (PAT), and since it is a cross-sectional study, only the main variable evaluated by the instrument will be described: psychosocial risk in pediatric health.

Conceptual Definition: Those dispositional variables (economic, social and structural factors for the care of pediatric cancer patients, among others) and functional variables (stress, anxiety, among others) specific that can influence the adaptation of primary caregivers to the treatment of their tutor.

Operational Definition:

The responses issued by the informal primary caregivers of pediatric cancer patients when answering the Psychosocial Risk Tool already translated and adapted for them. Considering the factors that make up this instrument:

* Family structure and resources
* Family problems
* Social support
* Children's problems
* Acute stress
* Sibling Problems

According to the characteristics of psychometric studies on instruments that are in another language, which require translation and adaptation, these are composed of four stages:

* Translation of the inventory from the original language (English - Spanish).
* Reverse translation of the inventory into the original language (Spanish - English).
* Validity of content, by expert judges.
* Piloting and obtaining the construct validity and reliability indices of the inventory with the target sample.

The four stages that will be carried out will be described below, following the recommendations suggested by the methodological guidelines of the International Test Commission (ICT) [60] and since it is a psychological assessment instrument, the recommendations of the consensus standards for the selection of health measurement instruments (COSMIN) [62] were added to the methodology to achieve this objective. The procedures of these stages will be described in the corresponding sections and in the procedure.

Sampling.

For translation, reverse translation and expert judging:

A non-probabilistic sampling will be used at convenience and 5 experts in pediatric oncological clinical psychology will be chosen, as proposed by Ato et al.

For the piloting of the translated and validated version:

A non-probabilistic convenience sampling will be used, according to the proposal of Streiner et al. , where it is recommended to select 10 individuals with characteristics similar to those of the target population.

For the collection of data to obtain the validity and reliability of the inventory:

Non-probabilistic convenience sampling will be used, which does not necessarily require random sample selection.

Sample Calculation

For the collection of data to obtain the validity and reliability of the inventory:

The sample size will be calculated by means of a mean difference test between two independent means (two groups) with a t-distribution, where it will be considered with an alpha equal to 0.05, α probability error to 0.05, effect size d=0.5, a statistical power equal to 0.95 and an assignment of two groups. considering a two-tailed distribution. Based on these values, a total sample size of 236 informal primary caregivers was calculated, where 118 participants will be collected for each center. The calculation was performed using g*power software 3.1.9.7.

Ethical aspects The research procedures will be carried out based on the Belmont Report, since the corresponding instruments will be applied, based on the informed consent that will be delivered to the participants (informal primary caregivers), where aspects such as the objectives, procedures, benefits of the study and the access they will have to the results will be found [66].

During the study, the informal primary caregivers will be asked for sensitive data on the minor; therefore, the generation of transparency and protection of information will be sought when making a plan for data processing, because it seeks to safeguard the ARCO rights of the participants, since they are the set of rights through which the Organic Law on the Protection of Personal Data, It guarantees individuals the power of control over their personal data, which will be described in the section on data processing [70]. The University of Kentucky's Informed Consent Checklist will be applied to safeguard the bioethical principles of participants [71].

This study is cross-sectional, which suggests a low risk; however, due to the nature of the instrument it can generate emotional responses in informal primary caregivers, to manage this situation, the team has assigned Alejandro Hernández Posadas, who has clinical experience in crisis intervention and belongs to the Association for the Help of Children with Cancer: "Aquí Nadie se Rinde I.A.P", so it has enough experience and knowledge to care for these caregivers. Your cell phone number will be provided to parents and will be available 24/7. This number is described in the informed consent that is sent to the committees of this institute for review and that will later be delivered to the parents.

If the research team identifies a moderate to severe mental health problem in caregivers, they will be given containment at first and then provide information about specialized public institutions near their place of origin where they can go for help, since visits to the institute are no longer frequent due to the pandemic.

Materials and Instruments The psychometric characteristics of the original inventory Psychosocial Assessment Tool (PAT) are described [72].

For Spanish-English translation A translation format has been created for 68 items, answer options and instructions for the Spanish version of an inventory.

For back-translation (English-Spanish) A translation format for the English version of the inventory, which includes instructions, response options and 68 items, has been developed and is based on the first translation.

For expert judging With the options of translation and inverted translation, taking care of the semantic content, the versions of the items that were best represented were obtained and modifications were made to the wording to adapt them to primary caregivers of pediatric cancer patients, so that they could design the judging format so that they could be evaluated by 10 expert psychologists and obtain a version close to the final one.

For piloting with the target population and collecting data on the validity and reliability of the inventory:

A document will be written in word office with: cover page, invitation letter, brief description of the characteristics, background of the inventory and its objective, as well as the privacy notice and informed consent.

All the instruments necessary for this study have the advantage of having dichotomous responses, and they will also be captured by the health professional in the institution (), with this they can be captured through electronic platforms such as Survey Monkey.

The reagents that will be captured on the platform will be:

• 68 questions from the Psychosocial Risk Tool, in its Mexican version for informal primary caregivers of childhood cancer survivors.

By capturing them, a link will be generated that can be shared with caregivers and from any electronic device (cell phone, tablet, laptop, desktop computer, etc.) they will be able to answer it.

Procedure The first three sections have been carried out and are described below. For Spanish-English translation A format was created to translate from English to Spanish and a professional translator was sought, who was a native Mexican and who had also had experience in an English-speaking culture, specifically in the United States. The aim was for the translator to be able to understand the intention behind each item and to maintain the psychological sense of the corresponding dimensions of the inventory and each item. The translator will be in charge of translating the 68 items, the instructions and the four answer options corresponding to each section. After the translation, a quantitative analysis of the direct translation will be carried out, with the help of an expert psychologist and the translator, to choose the most suitable translation.

For English-Spanish back-translation. A reverse translation format (English-Spanish) was created using the pre-translation of the items, instructions, and answer options. An expert translator in English and Spanish who is also a psychologist and is a native of an English-speaking country (United States, Texas) was hired. This translator was unaware of the inventory and was in charge of translating the Spanish version, instructions, answer options and the 68 items. The translated version was compared with the original version of the inventory to identify concordance and determine the best version of each item for the target population.

For expert judging Once the semantic equivalence of the items was achieved and the wording was adjusted so that the inventory was appropriate for informal primary caregivers of pediatric cancer patients, a format was designed for experts to assess the content validity of the inventory. 10 psychologists with master's degrees specialized in psycho-oncology, behavioral medicine, and child psychology were selected to evaluate the psychometric quality, theoretical content, and validity of each of the 68 items. They were provided with information on the objective of the research, the defined construct and the dimensions that compose it, and they were given a judging form to evaluate the relevance, writing, appropriate language for the population, theoretical validity, criterion validity and content validity of each of the 68 items, answer options and instructions. In addition, they were asked to comment on possible adaptations or changes in the wording of these elements to make them more understandable to the target population.

For piloting with the target population In the waiting room, informal primary caregivers who meet the criteria set out to participate in the study will be identified and explained the purpose of the research and the importance of their participation in the pilot evaluation. In addition, they will be assured that they will have the necessary resources to respond to the questionnaire and will be guaranteed the confidentiality of the information provided, which will only be used for statistical and scientific purposes. Since caregivers may be in different situations, several options will be offered to obtain informed consent and the document will be required to be signed by the caregivers and two witnesses, who will confirm that participation was not compelled and that there are no hidden interests.

Then, the health professional will apply the instrument through the "survey monkey" platform and the answers will be automatically sent to a database to which only the research team will have access. It will be verified that all the items in the battery have been answered. Caregivers' suggestions on items, instructions, response options, and the application process will be qualitatively analyzed. Based on these analyses, adjustments will be made and the final electronic version of the battery will be obtained for use.

For data collection to obtain the validity and reliability of the scale:

Informal primary caregivers will be selected in the waiting room using the inclusion and exclusion criteria for study participants. Once selected, the purpose of the research will be explained to the CPIs, the importance of their participation in the pilot evaluation, and it will be ensured that they have the necessary resources to respond to the questionnaire (computer, tablet or phone with a program that allows the editing of the document). In addition, the confidentiality of the information provided will be ensured and its use will only be for statistical and scientific purposes. Since caregivers may be in different contexts, different options will be offered to obtain informed consent. These documents must be signed together with two witnesses who can attest that the participation was not coerced and that there are no hidden interests. It is important to note that, as it is a multicenter study, in which the Federico Gómez Children's Hospital of Mexico and the National Institute of Pediatrics will participate; therefore, the instrument will be applied at the same time, for a period of time of two months, through the "survey monkey" platform by the health professional, the Survey Monkey program automatically sends the responses to a database that only the research team has access, it will be checked that the battery has been completed in its entirety. It is indicated that, if there are any side effects from the application of the scale, a telephone number will be provided to provide crisis care, in case the caregiver needs it. Likewise, they are told that they will be notified about the results obtained and it is important that they remember the folio number assigned by the program. In the event that any mental health problems are detected, information will be provided on nearby places to receive care, so that the parent is informed about where to go if necessary Data analysis for validation For the expert judging The indices of relevance, writing, and appropriate language for the population were obtained, in order to obtain the apparent validity and content validity of each of the 68 items, through the evaluation carried out by experts. With these results, the reliability of each characteristic was calculated as an independent category, using the corresponding coefficient. Descriptive statistics were used to analyze the central tendency frequencies of the participants' characteristics.

Data analysis for instrument validation Feasibility: This section will record the time it took participants to complete the scale, the difficulties they faced in answering questions, and the number of missing values (patients who did not respond) for each question. The items will be analyzed by calculating the frequency of each response category in each of them, as well as the rate of missing responses for each item. The effects of "floor" and "ceiling" will also be analyzed, both in each item and in the global questionnaire.

Reliability: Reliability will be assessed by calculating the Kuder-Richardson 20 coefficient (KR20) to determine internal consistency.

Validity:

a) Construct: Structural or construct validity will be evaluated using exploratory factor analysis. The common factor model, the minimum waste extraction method and the Oblimin rotation (if possible) will be used. The K1 rule (eigenvalues greater than one) and the Cattell screen test will be used to determine the number of factors in the solution. In addition, a confirmatory factor analysis will be performed to confirm the original structure, assuming the presence of a single factor in which all items will be loaded.

Conflict of interest:

This research has been funded by Aquí Nadie se Rinde IAP

ELIGIBILITY:
Inclusion Criteria:

* Informal primary caregivers of pediatric cancer patients, who verbally state that they have assumed responsibility for care from diagnosis to survival.
* Informal primary caregivers of pediatric cancer patients over 18 years of age.
* Informal primary caregivers of pediatric cancer patients who can read and write.
* Informal primary caregivers of pediatric cancer patients who are receiving chemotherapy and/or radiation therapy.
* Informal primary caregivers of pediatric cancer patients who agree to participate in the study.

Exclusion Criteria:

* Informal primary secondary caregivers of pediatric cancer patients.
* Informal primary caregivers of pediatric cancer patients who have participated in the piloting of the study.
* Informal primary caregivers of pediatric cancer patients who are receiving palliative care treatment.
* Informal primary caregivers of pediatric cancer patients who are in remission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants:
  For Spanish-English translation and back-translation According to the guidelines of the International Test Commission [63], the participation of an experienced native Mexican translator who is or has been immersed in the English-speaking culture will be required.
  On the other hand, for translation from English to Spanish, a native translator from an English-speaking country with experience who is immersed in Mexican culture will be required for translation from Spanish to English.
  For expert judging The participation of 10 psychologists who are experts in the following areas (psycho-oncology, health psychology and behavioural medicine with postgraduate qualifications for expert judging) will be required.
  For the piloting of the translated and validated version:
  10 informal primary caregivers of pediatric cancer patients who come to the National Institute of Pediatrics will be necessary.
Sampling Method: Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Psychosocial Assessment Tool | 3 months
  The PAT is a brief report for informal primary caregivers that assesses family psychosocial risk based on a families' ecological social model. This model assesses psychosocial risks throughout the child's social environment and generates seven subscale scores, such as Family Structure/Resources, Social Support, Children's Problems, Sibling Problems, Family Problems, Stress Reactions, and Family Beliefs [61]. The total score, which ranges from 0 to 7, is assigned to the PPPHM (Kazak, 2006) with three risk levels: universal (<1.00), specific (1.00 and 2.00) and clinical (>2.00). To translate the PAT into Spanish, methods that met or exceeded the guidelines of Holmbeck and Devine were used. First, the PAT was independently translated and back-translated by two native Spanish-speaking psychologists. Then, an independent native Spanish speaker reviewed it and consulted with a certified translator.

CONTACTS AND LOCATIONS:
Locations (1):
- Aquí Nadie se Rinde I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] References: 1. Foreman KJ, Marquez N, Dolgert A, Fukutaki K, Fullman N, McGaughey M, et al. Forecasting life expectancy, years of life lost, and all-cause and cause-specific mortality for 250 causes of death: reference and alternative scenarios for 2016-40 for 195 countries and territories. Lancet. 2018; 392(10159):2052-90. https://pubmed.ncbi.nlm.nih.gov/30340847/ 2. Bray F, Jemal A, Grey N, Ferlay J, Forman D. Global cancer transitions according to the Human Development Index (2008-2030): a population-based study. Lancet Oncol. 2012; 13(8):790-801. https://pubmed.ncbi.nlm.nih.gov/22658655/ 3. CP W, E W, BW S. World Cancer Report: Cancer Research for Cancer Prevention [Internet]. [citado 19 de marzo de 2023]. Disponible en: https://publications.iarc.fr/Non-Series-Publications/World-Cancer-Reports/World-Cancer-Report-Cancer-Research-For-Cancer-Prevention-2020 4. Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, et al. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. mayo de 2021; 71(3):209-49. https://pubmed.ncbi.nlm.nih.gov/33538338/ 5. Home | Sustainable Development [Internet]. [cited 2023 March 19]. Available in: https://sdgs-un-org.pbidi.unam.mx:2443/ 6. NCD Countdown 2030 collaborators. NCD Countdown 2030: worldwide trends in non-communicable disease mortality and progress towards Sustainable Development Goal target 3.4. Lancet. 2018; 392(10152):1072-88. https://www.thelancet.com/pb-assets/Lancet/hubs/ncd/NCDCountdown2030_Summary_FINAL-1537452913640.PDF 7. NCD Countdown 2030 collaborators. NCD Countdown 2030: pathways to achieving Sustainable Development Goal target 3.4. Lancet. 2020; 396(10255):918-34. https://www.thelancet.com/journals/lancet/article/PIIS0140-6736(18)31992-5/fulltext 8. Kuderer NM, Choueiri TK, Shah DP, Shyr Y, Rubinstein SM, Rivera DR, et al. Clinical impact of COVID-19 on patients with cancer (CCC19): a cohort study. Lancet. 2020